CLINICAL TRIAL: NCT02119429
Title: The Effect of Pumpkin Seed Oil Supplementation on Blood Pressure in Premenopausal Women
Brief Title: Pumpkin Seed Oil Supplementation in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17411a
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-12

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Pre-menopausal; Supplementation
MeSH Terms: interventions — wheat germ oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wheat Germ Oil (Placebo Comparator): Participants will be instructed to consume 2 wheat germ oil capsules ,2g, per day for 12 weeks.
  Interventions: Dietary Supplement: Wheat Germ Oil
- Pumpkin Seed Oil (Experimental): Participants will be instructed to consume 2 pumpkin seed oil capsules ,2g, per day for 12 weeks
  Interventions: Dietary Supplement: Pumpkin Seed Oil

INTERVENTIONS:
Dietary Supplement: Pumpkin Seed Oil — 2 grams per day, everyday for 12 weeks.
  Arms: Pumpkin Seed Oil
Dietary Supplement: Wheat Germ Oil — 2 grams per day, everyday for 12 weeks.
  Arms: Wheat Germ Oil

SUMMARY:
The purpose of this study is to determine whether or not there is an effect of pumpkin seed oil supplementation, 2 grams per day, on blood pressure (systolic and diastolic) in premenopausal women.

DETAILED DESCRIPTION:
The research study will be conducted over a 12-week period. Overall, each participant will meet with the researcher three times. During the first visit, after the participant has signed the consent form, their blood pressure will be taken with a digital blood pressure monitor. If her systolic blood pressure is greater than 140 mmHg or her diastolic blood pressure is greater than 90 mmHg, she will not be eligible to take part in this study. If the participant is able to take part in this study, she will be given a code number to protect confidentiality and randomly assigned to one of two groups, Group I or Group II. The participant will then be asked to state their age, ethnicity, menopausal status, and whether or not they are taking oral contraceptives. Next, height and weight will be taken with an instrument called a Health-O-Meter. Body mass index (BMI) and percent body fat will be calculated using an instrument called a Body Composition Analyzer. After all measurements are taken, participants will be given instructions on how to keep a 3-day diet and supplement diary. A booklet will be provided to help them record their diet for two nonconsecutive week days and one weekend day. The 3-day diet and supplement diary is to be completed during the week between the first and second session with the researcher. During this session the participant will be asked to complete a food frequency questionnaire to help the researcher asses the phytoestrogen content of her diet. At the end of the first session, the researcher will schedule a second session with the participant.

The second session will take place one week after the first session. During the second session, measurements taken will be height, weight, BMI, percent body fat, and blood pressure. Participants will be asked to return the 3-day diet and supplement diary to the researcher. The researcher will review the diary and ask questions to clarify foods recorded. The participant will then be asked to complete a physical activity questionnaire. Next, supplements will be distributed. The participants will not have knowledge of which group they are assigned to. Group I will receive 168 capsules, each capsule containing 1 gram of wheat germ oil, in two pill bottles. One bottle will contain 100 capsules; the second bottle will contain 68 capsules. Group II will receive 168 capsules, each capsule containing 1 gram of pumpkin seed oil, in two pill bottles. One bottle will contain 100 capsules; the second bottle will contain 68 capsules. Participants will be instructed to take 2 capsules per day, every day for 12 weeks. Two capsules per day are equal to approximately a ½ teaspoon or 18 kilocalories. It does not matter if they choose to take each capsule at the same time or at different times during the day. To help remind participants to take their supplements each day, they will receive a 7 day pill organizer and a daily check list. At this session, participants will receive a second 3-day diet and supplement diary that is to be completed one week before the final session. At the end of the second session, the researcher will schedule the final session with the participant.

The third and final session will take place 12 weeks after the initial session. Measurements taken during the final session will be height, weight, BMI, percent body fat, and blood pressure. The participant will be asked to complete a food frequency questionnaire identical the questionnaire filled out during the first session with the researcher. Participant will be asked to return their 3-day diet and supplement diary, daily check list, pill organizer, 2 pill bottles, and any unused supplements. After completion of the study the participant will receive a $20 Target gift card at this session.

A potential risk of this study includes loss of confidentiality. Confidentiality will be maintained by the use of code numbers rather than names on data containing documents. Digital data analyses will be done using only code numbers and not identifiable data. Data recorded on paper containing identifiable and non-identifiable participant information (consent forms, data collection forms, 3-day diet and supplement diaries, physical activity questionnaires, food frequency questionnaires, and participant daily checklists) will be kept in a locked cabinet in Room 10132B in the Texas Woman's University, Houston Office of Research.

Another potential risk of this study may be that the participant's normal schedule is disrupted by coming to the Texas Woman's University, Houston campus. To minimize this risk, sessions will be scheduled with the researcher in advance Monday through Friday, from 8 a.m. to 5 p.m. to accommodate the participant's schedule.

ELIGIBILITY:
Inclusion Criteria:

* Read, speak, and write English
* Premenopausal

Exclusion Criteria:

* Consuming estrogen supplements
* Taking hypertensive blood pressure medication
* Consuming pumpkin seed oil supplements
* Consuming pumpkin seeds more than once a month
* Wheat allergy or gluten intolerance
* Blood pressure > 140/90 mmHg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Systolic Blood Pressure at 12 weeks | Baseline, 12 weeks
Change From Baseline Diastolic Blood Pressure at 12 weeks | Baseline, 12 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline
  BMI is an important measurement to record because an increase in weight may be accompanied by an increase in blood pressure.
Percent Body Fat | Baseline
  Percent body fat is an important measurement to record because an increase in body fat may be accompanied by an increase in blood pressure.
Nutrient content of diet | Baseline
  Participants will be given instructions on how to keep a 3-day diet and supplement diary. A booklet will be provided to help them record their diet for two nonconsecutive week days and one weekend day. Diet will then be analyzed using Minnesota Nutrition Data System for calories, carbohydrate, protein, fat, vitamins, minerals, and phytoestrogen content.
Phytoestrogen content of diet | Baseline
  A food frequency questionnaire will be given to each participants to assess the phytoestrogen content of her diet.
Activity Level | Baseline
  The purpose of the physical activity questionnaire is to establish each participant's activity level because physical activity level may have an effect on blood pressure.
Body Mass Index (BMI) | 12 weeks
  BMI is an important measurement to record because an increase in weight may be accompanied by an increase in blood pressure.
Percent Body Fat | 12 weeks
  Percent body fat is an important measurement to record because an increase in body fat may be accompanied by an increase in blood pressure.
Nutrient content of diet | 12 weeks
  Participants will be given instructions on how to keep a 3-day diet and supplement diary. A booklet will be provided to help them record their diet for two nonconsecutive week days and one weekend day. Diet will then be analyzed using Minnesota Nutrition Data System for calories, carbohydrate, protein, fat, vitamins, minerals, and phytoestrogen content.
Phytoestrogen content of diet | 12 weeks
  A food frequency questionnaire will be given to each participants to assess the phytoestrogen content of her diet.
Activity Level | 12 weeks
  The purpose of the physical activity questionnaire is to establish each participant's activity level because physical activity level may have an effect on blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha L Caudill, BS, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Institute of Health Sciences- Houston Center, Houston, Texas, United States